CLINICAL TRIAL: NCT04357769
Title: A Study of Perceived Distress and Psychological Burden in Patients Suffering From Severe Mental Diseases During the COVID-19 Pandemic in Italy
Brief Title: COVID-19 Pandemic Burden in Severe Mental Disease Patients
Acronym: PsyCOVID
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Felice Iasevoli, Associate Professor of Psychiatry, Federico II University
Other Study IDs: 152/20
Record Dates: First submitted 2020-04-16; First posted 2020-04-22 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Psychological Distress; COVID; Severe Mental Disorder
MeSH Terms: conditions — Mental Disorders | interventions — Perceived Stress Scale; Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients: Individuals aged 18-70 years with a diagnosis of severe mental disorder (schizophrenia or psychosis spectrum disorder; bipolar disorder; major depressive disorder) who were in a condition of psychopathological compensation, had their last clinical evaluation at the University of Naples Federico II outpatient unit of Psychiatry during January-February 2020, were not positive or suspected positive for COVID-19, and were under strict quarantine
  Interventions: Other: PSS (Perceived Stress Scale); Other: GAD-7 (7-item Generalized Anxiety Disorder); Other: PHQ-9 (9-item Patient Health Questionnaire); Other: SPEQ (Specific Psychotic Experiences Questionnaire) - Paranoia and Grandiosity Subscales
- Controls (General Population): Individuals aged 18-70 years who had not a psychiatric condition nor were positive or suspected positive for COVID-19 and were under strict quarantine (e.g. not getting out for work)
  Interventions: Other: PSS (Perceived Stress Scale); Other: GAD-7 (7-item Generalized Anxiety Disorder); Other: PHQ-9 (9-item Patient Health Questionnaire); Other: SPEQ (Specific Psychotic Experiences Questionnaire) - Paranoia and Grandiosity Subscales
- First-degree Relatives: Individuals aged 18-70 years who were first-degree relatives and caregivers of an individual included in the Patients group, who had not a psychiatric condition nor were positive or suspected positive for COVID-19 and were under strict quarantine
  Interventions: Other: PSS (Perceived Stress Scale); Other: GAD-7 (7-item Generalized Anxiety Disorder); Other: PHQ-9 (9-item Patient Health Questionnaire); Other: SPEQ (Specific Psychotic Experiences Questionnaire) - Paranoia and Grandiosity Subscales; Other: Zaritt Burden Interview

INTERVENTIONS:
Other: PSS (Perceived Stress Scale) — Self-administered scale for the evaluation of the stress perceived by the subject in the last weeks
Other: GAD-7 (7-item Generalized Anxiety Disorder) — Self-administered scale for the evaluation of anxiety symptoms in the last weeks
Other: PHQ-9 (9-item Patient Health Questionnaire) — Self-administered scale for the evaluation of depressive symptoms in the last weeks
Other: SPEQ (Specific Psychotic Experiences Questionnaire) - Paranoia and Grandiosity Subscales — Self-administered scale for the evaluation of sub-threshold psychotic symptoms in the last weeks
Other: Zaritt Burden Interview — Self-administered scale for the evaluation of severe mental disorder patients' caregiver burden
  Groups: First-degree Relatives

SUMMARY:
Despite being originated in Wuhan, in the China mainland region of the Hubei, Italy has been the hardest-hit country in the world by the COVID-19 pandemic during the month of March.

Due to the uncontrollable spread of the contagion, the Italian Government has been forced to impose a series of restrictions and social distancing measures, culminating in the extension of lockdown to the entire Italian territory on March 8th.

During this period, the general population has been overwhelmed by feelings of worry, anxiety, and discomfort. The discomfort is reinforced by the lengthening of the lockdown, to the point that it may be considered as a mass model of chronic or subchronic mild stress.

The predictable effects of this stress on mental health have already been claimed, Post-traumatic symptoms were found in 7% among 285 Wuhan and surrounding cities' residents during the COVID-19 outbreak. A recent survey in the Italian general population reported similar outcomes.

In this context, the psychic conditions of the most fragile ones, i.e. those already affected by a severe mental disorder, represent a major concern. Having a history of psychiatric illness is regarded as one of the most relevant predictors of a negative psychological impact of quarantine. Patients with severe mental disorders may be among the hardest hit subjects, as they may be more vulnerable by the COVID-19 outbreak for a series of clinical and psychological factors. In the Italian context, the vulnerability of these patients may be increased by the lockdown of mental health services as a consequence of mass quarantine and optimization of health resources toward action to contrast COVID-19-related sanitary emergencies.

Despite several reports investigated the psychological effects of COVID-19 pandemic on health-care workers, COVID-19 affected people, or the general population, at the moment, no study has investigated the effects of the distress caused by fear of contagion and mass quarantine on severe mental disorder patients. The present study aimed at providing a first evaluation of anxiety, depressive, stress-related symptoms in these patients.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 Diagnosis of Schizophrenia or Psychosis Spectrum; Bipolar Disorder; REcurrent Major Depressive Disorder
* Linguistic and cognitive ability to complete the rating scales
* Written informed consent
* Psychopathological compensation at last clinical evaluation on January-February 2020

Exclusion Criteria:

* SARS-CoV-2 positive, suspected positive, or in recent close contact with positive ones
* Not under strict quarantine, due to work reasons or to any other reason allowing to overcome quarantine
* Current or recent hospitalization (i.e. on March-April), for any reason
* Intellectual disability
* Psychiatric disturbances secondary to general medical conditions or substances
* Serious medical conditions with infaust prognosis or severely affecting the quality of life
* Living in Northern Italy

Adjunctive Exclusion Criteria for the General Population and Caregivers:

* Psychiatric Disorder, of any type

Adjunctive Exclusion Criteria for the General Population:

* First degree relative or caregiver of a psychiatric patient

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All subjects included in the study should have been under mass quarantine in the last month and should have been exposed to similar distressing factors during the SARS-CoV-2 outbreak in Italy
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) outcome | 10 days
  Significant differences among groups in the mean Perceived Stress Scale (PSS) score, which measures the stress severity perceived by the subjects in the last month. The scale is constituted by 10 items that are self-rated by the subject on a 0-4 Likert scale. The scale minimum total score is 0, the maximum is 40. Higher total scores indicate a worse outcome

SECONDARY OUTCOMES:
Generalized Anxiety Disorder (GAD-7) scale outcome | 10 days
  Significant differences among groups in the mean Generalized Anxiety Disorder (GAD-7) scale score, which measures anxiety symptoms' severity in the last two weeks. The scale is constituted by 7 items that are self-rated by the subject on a 0-3 Likert scale. The scale minimum total score is 0, the maximum is 21. Higher total scores indicate a worse outcome
Patient Health Questionnaire (PHQ-9) scale outcome | 10 days
  Significant differences among groups in the mean Patient Health Questionnaire (PHQ-9) scale score, which measures depressive symptoms' severity in the last two weeks. The scale is constituted by 9 items that are self-rated by the subject on a 0-3 Likert scale. The scale minimum total score is 0, the maximum is 21. Higher total scores indicate a worse outcome
Specific Psychotic Experiences Questionnaire (SPEQ) - Paranoia subscale outcome | 10 days
  Significant differences among groups in the mean Specific Psychotic Experiences Questionnaire (SPEQ) - Paranoia subscale score. The SPEQ scale is designed for the assessment of current sub-threshold psychotic symptoms in multiple domains. The Paranoia subscale measures persecutory/reference ideas and is constituted by 15 items that are self-rated by the subject on a 0-5 Likert scale. The subscale minimum total score is 0, the maximum is 75. Higher total scores indicate a worse outcome
Specific Psychotic Experiences Questionnaire (SPEQ) - Grandiosity subscale outcome | 10 days
  Significant differences among groups in the mean Specific Psychotic Experiences Questionnaire (SPEQ) - Grandiosity subscale score. The Grandiosity subscale measures grandiosity/megalomaniac ideas and is constituted by 8 items that are self-rated by the subject on a 0-3 Likert scale. The subscale minimum total score is 0, the maximum is 24. Higher total scores indicate a worse outcome
Caregiver Burden | 10 days
  Significant correlations between mean Zarit Burden Interview (ZBI) and mean scores on the Perceived Stress Scale (PSS). The ZBI is designed for the assessment of caregiver burden. The scale is constituted by 22 items that are self-rated by the subject on a 0-4 Likert scale. The scale minimum total score is 0, the maximum is 88. Higher total scores indicate a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples "Federico II", Napoli, Italy

IPD SHARING:
Plan to Share IPD: Undecided